CLINICAL TRIAL: NCT01174004
Title: A Multi-Center, Placebo-Controlled, Double-Blind Trial to Examine the Safety and Efficacy of Pimavanserin in the Treatment of Psychosis in Parkinson's Disease
Brief Title: A Study of the Safety and Efficacy of Pimavanserin in Patients With Parkinson's Disease Psychosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-103-020
Record Dates: First submitted 2010-07-30; First posted 2010-08-03 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Parkinson's Disease Psychosis
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): pimavanserin tartrate, 40 mg, tablet, once daily by mouth for 6 weeks
  Interventions: Drug: pimavanserin tartrate
- 2 (Placebo Comparator): placebo, tablet, once daily by mouth for 6 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pimavanserin tartrate — pimavanserin tartrate, 40 mg, tablet, once daily by mouth for 6 weeks
  Other Names: ACP-103
  Arms: 1
Drug: placebo — placebo, tablet, once daily by mouth for 6 weeks
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of 40 mg pimavanserin compared to placebo in patients with Parkinson's disease psychosis (PDP).

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of Parkinson's disease with a minimum duration of 1 year
* Presence of visual and/or auditory hallucinations, and/or delusions, occurring during the four weeks prior to study screening
* Psychotic symptoms must have developed after Parkinson's disease diagnosis was established
* Subjects that are on anti-Parkinson's medication must be on a stable dose for 1 month prior to Study Day 1 (Baseline) and during the trial
* Subject that has received stereotaxic surgery for subthalamic nucleus deep brain stimulation must be at least 6 months post surgery and the stimulator settings must have been stable for at least 1 month prior to Study Day 1 (Baseline) and must remain stable during the trial
* The subject is willing and able to provide consent
* Caregiver is willing and able to accompany the subject to all visits
* Subject and caregiver are willing and able to adequately communicate in English for the purposes of the primary assessment

Exclusion Criteria:

* Subject has a history of significant psychotic disorders prior to or concomitantly with the diagnosis of Parkinson's disease including, but not limited to, schizophrenia or bipolar disorder
* Subject has received previous ablative stereotaxic surgery (i.e., pallidotomy and thalamotomy) to treat Parkinson's disease
* Subject has current evidence of a serious and or unstable cardiovascular, respiratory, gastrointestinal, renal, hematologic or other medical disorder
* Subject has had a myocardial infarction in last six months
* Subject has any surgery planned during the screening, treatment or follow-up periods

Patients will be evaluated at screening to ensure that all criteria for study participation are met. These evaluations will include specific measures of psychosis severity, delirium, dementia, cardiovascular condition, and pregnancy status. Patients may be excluded from the study based on these assessments (and specifically if it is determined that their baseline health and psychiatric condition do not meet all protocol-specified entry criteria).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2010-07; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (61):
  - Gilbert, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Carson, California
  - Fountain Valley, California
  - Fresno, California
  - Fullerton, California
  - Irvine, California
  - La Habra, California
  - La Jolla, California
  - Loma Linda, California
  - Oxnard, California
  - Pasadena, California
  - Reseda, California
  - Sunnyvale, California
  - Ventura, California
  - Danbury, Connecticut
  - Boca Raton, Florida
  - Bradenton, Florida
  - Naples, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Panama City, Florida
  - Port Charlotte, Florida
  - St. Petersburg, Florida
  - Augusta, Georgia
  - Decatur, Georgia
  - Elk Grove Village, Illinois
  - Glenview, Illinois
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Scarborough, Maine
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Novi, Michigan
  - Roseville, Michigan
  - Traverse City, Michigan
  - Flowood, Mississippi
  - St Louis, Missouri
  - Missoula, Montana
  - Toms River, New Jersey
  - Albany, New York
  - Commack, New York
  - Kingston, New York
  - New York, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Greensburg, Pennsylvania
  - Providence, Rhode Island
  - Brentwood, Tennessee
  - Houston, Texas
  - Salt Lake City, Utah
  - Alexandria, Virginia
  - Roanoke, Virginia
  - Virginia Beach, Virginia
  - Milwaukee, Wisconsin
- Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Cummings J, Isaacson S, Mills R, Williams H, Chi-Burris K, Corbett A, Dhall R, Ballard C. Pimavanserin for patients with Parkinson's disease psychosis: a randomised, placebo-controlled phase 3 trial. Lancet. 2014 Feb 8;383(9916):533-40. doi: 10.1016/S0140-6736(13)62106-6. Epub 2013 Nov 1. PMID 24183563

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablet, once daily by mouth, 6 weeks
- Pimavanserin 40 mg: Pimavanserin tartrate (ACP-103), 40 mg, tablet, once daily by mouth, 6 weeks
Period: Overall Study
Arm/Group | Placebo | Pimavanserin 40 mg
Started | 94 | 105
Completed | 87 | 89
Not Completed | 7 | 16
Not completed — Adverse Event | 2 | 10
Not completed — Withdrawal by Subject | 2 | 3
Not completed — At Discretion of Sponsor | 2 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pimavanserin 40 mg | Total
Number analyzed (Participants) | 94 | 104 | 198
Age, Categorical [Count of Participants; unit: Participants] — Safety Analysis Set
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 11 | 12 | 23
    >=65 years | 83 | 92 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (8.03) | 72.6 (6.49) | 72.7 (7.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 34 | 72
  Male | 56 | 70 | 126
Region of Enrollment [Number; unit: participants]
  United States | 92 | 101 | 193
  Canada | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Antipsychotic Efficacy
Description: Antipsychotic Efficacy was defined as a decrease in the severity and/or frequency of hallucinations and/or delusions. This is measured as the change from baseline (Day 1) to Day 43 in the Scale for the Assessment of Positive Symptoms 9-item sum score for Parkinson's Disease (SAPS-PD). The possible total score is 0 to 45 and a negative change in score indicates improvement.
  Analysis Method: Mixed Model Repeated Measures (MMRM)
Time Frame: Each study visit (i.e. Days 1, 15, 29 and 43)
Population: This is the "Intent to Treat" population, defined as patients who received at least one dose of study drug and had both the baseline SAPS assessment and at least one post-baseline SAPS assessment collected no later than 3 days after the last dose date.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on the SAPS-PD scale
Arm/Group | Placebo | Pimavanserin 40 mg
Number analyzed (Participants) | 90 | 95
Score on the SAPS-PD scale
  Change from Baseline | -2.73 [-4.05 to -1.42] | -5.79 [-7.09 to -4.49]
  Difference of Least Squares Mean versus Placebo | NA [NA to NA] — Calculation is a comparison of active arm versus placebo. | -3.06 [-4.91 to -1.20]

2. Secondary Outcome: Motor Symptoms Change From Baseline (Negative = Improvement)
Description: Motor symptoms were measured using the change from baseline to Day 43 in the combined score of the Unified Parkinson's Disease Rating Scale (UPDRS) Part II (Activities of Daily Living) and Part III (Motor Examination). The possible total score is 0 to 160 and a negative change in score indicates improvement.
  Analysis Method: Analysis of Covariance (ANCOVA). The UPDRS Parts II+III score was analyzed by constructing 2-sided 95% confidence intervals (CIs) on the difference between the pimavanserin dose group and placebo mean change from baseline. Non-inferiority was concluded if the upper limit of the CI was less than or equal to 5.
Time Frame: Study Days 1 and 43
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on the UPDRS-II+III
Arm/Group | Placebo | Pimavanserin 40 mg
Number analyzed (Participants) | 90 | 95
Score on the UPDRS-II+III
  Change from Baseline | -1.69 [-3.43 to 0.05] | -1.40 [-3.10 to 0.30]
  Difference of Least Squares Mean versus Placebo | NA [NA to NA] — Calculation is a comparison of active arm versus placebo. | 0.29 [-2.14 to 2.72]

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: From the time the informed consent was signed, adverse events were recorded in the subject's source documents and entered into the appropriate eCRF pages at the Screening visit, at visits on Study Days 1, 15, 29, 43 and Day 71 or 4 weeks after the last dose for subjects who do not continue into the open-label, extension protocol.
Arm/Group | Placebo | Pimavanserin 40 mg
Serious Adverse Events (participants affected / at risk) | 4/94 | 11/104
Other Adverse Events (participants affected / at risk) | 31/94 | 41/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=94) | Pimavanserin 40 mg (N=104)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=94) | Pimavanserin 40 mg (N=104)
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (7)
Edema peripheral (General disorders) | 3 (3) | 7 (7)
Urinary tract infection (Infections and infestations) | 11 (12) | 14 (16)
Fall (Injury, poisoning and procedural complications) | 8 (9) | 11 (14)
Confusional state (Nervous system disorders) | 3 (4) | 6 (6)
Headache (Nervous system disorders) | 5 (5) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment.